CLINICAL TRIAL: NCT06310954
Title: The Efficacy of Ketogenic Diet in Treating Pediatric Intractable Epilepsy and Its Relationship With Changes in Inflammatory Markers
Brief Title: Ketogenic Diet in Pediatric Intractable Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-KY-012
Record Dates: First submitted 2024-01-22; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Epilepsy in Children; Epilepsy Intractable
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic Diet plus Conventional Treatment Group (Experimental): This arm of the trial explores the efficacy of an early initiation of the ketogenic diet in conjunction with conventional antiepileptic drugs (AEDs) for children with refractory epilepsy. The intervention aims to evaluate the impact on seizure frequency, and inflammatory markers, and identify patient characteristics predicting a better response to the ketogenic diet, to improve overall therapeutic response rates in refractory epilepsy.
  Interventions: Dietary Supplement: Early ketogenic diet combined with conventional pharmacotherapy.; Drug: Common diet combined with conventional pharmacotherapy
- Control Group: Conventional Treatment Group (Placebo Comparator): Participants in this arm will receive a standard diet without any ketogenic restrictions, alongside conventional antiepileptic drugs. This comparator aims to assess the standard care's efficacy against the experimental intervention, focusing on seizure control, inflammatory markers, and identifying patient characteristics associated with treatment responsiveness.
  Interventions: Dietary Supplement: Early ketogenic diet combined with conventional pharmacotherapy.; Drug: Common diet combined with conventional pharmacotherapy

INTERVENTIONS:
Dietary Supplement: Early ketogenic diet combined with conventional pharmacotherapy. — This arm of the trial explores the efficacy of an early initiation of the ketogenic diet in conjunction with conventional antiepileptic drugs (AEDs) for children with refractory epilepsy. The intervention aims to evaluate the impact on seizure frequency, and inflammatory markers, and identify patient characteristics predicting a better response to the ketogenic diet, to improve overall therapeutic response rates in refractory epilepsy.
Drug: Common diet combined with conventional pharmacotherapy — Participants in this arm will receive a standard diet without any ketogenic restrictions, alongside conventional antiepileptic drugs. This comparator aims to assess the standard care's efficacy against the experimental intervention, focusing on seizure control, and inflammatory markers, and identifying patient characteristics associated with treatment responsiveness.We know that drug information for registering clinical information is necessary, but our research design is to add ketogenic diets as a supplementary treatment plan when traditional drug treatment is ineffective. Therefore, in terms of specific drug selection, this is not absolutely the same. Depending on individual differences, the choice of drugs will also vary. Control the number of episodes, time, etc., and everyone uses different drugs. Therefore, we cannot decide on a single drug for comparison like traditional content.

SUMMARY:
This study aims to evaluate the efficacy of a ketogenic diet in treating pediatric intractable epilepsy and to explore its relationship with changes in inflammatory markers. The investigators plan to recruit 59 participants with intractable epilepsy, 39 of whom will receive a combination of ketogenic diet and conventional antiepileptic drugs, while 20 will receive only conventional drugs. The study will assess the impact of the ketogenic diet on epilepsy control and inflammatory markers, hoping to discover new treatment strategies.

DETAILED DESCRIPTION:
Evaluation index

1. Safety: Adverse events related to the ketogenic diet
2. Efficacy evaluation:

A. Primary efficacy indicators: brain electrical load index, epilepsy control response rate, inflammatory factor 34 (blood, cerebrospinal fluid) Secondary efficacy indicators: epilepsy seizure-free rate B. Inspection indicators: blood ketone, blood sugar, blood biochemistry testing, etc.; C. Use high-throughput methods to detect absolute counts of cerebrospinal fluid, serum inflammatory factors, and whole blood lymphocyte subpopulations before and after adding a ketogenic diet.

Observation indicators

1. Measurement of ketone body levels Monitor blood ketones (beta-hydroxybutyrate) and blood ketones. Recording time: Record three times a day during the baseline period; record the average blood ketone value at each subsequent follow-up observation.
2. Frequency of epileptic seizures The frequency of epileptic seizures was recorded daily during the start-up period.
3. Efficacy evaluation:

   Main efficacy indicators: epilepsy control response rate, seizure-free rate, inflammatory factor levels Epilepsy control response rate: defined as an absolute reduction of ≥50% in seizure frequency at follow-up compared with baseline

   =(No attack + Marked effect + Effective)/Total number of cases × 100%. Evaluation of seizure control: No seizures: seizures are completely relieved after treatment; Markedly effective: the number of seizures is reduced by ≥75% after treatment; Effective: the number of seizures is reduced by ≥50% after treatment; Ineffective: the number of seizures is reduced by <50% after treatment.

   Seizure-free rate: Seizures were completely controlled at follow-up. = No attack cases/Total number of cases × 100%
4. Safety evaluation Record various adverse events; biochemical monitoring (glucose and lipid metabolism and related tests); other tests: necessary tests according to the condition (blood gas analysis, B-ultrasound, etc.);
5. Physical development Monitor and record height and weight, and conduct physical development evaluation.
6. Cognitive-behavioral development assessment The baseline period, KD weeks 4, 12, and KD week 16 (at the end of the efficacy observation period) were evaluated and recorded using the Gesell score scale.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 12 years with a diagnosis of intractable epilepsy
* more than four seizures per month
* no metabolic diseases
* no severe liver or kidney dysfunction.

Exclusion Criteria:

* Fat metabolism or other metabolic diseases
* febrile or infectious periods
* contraindications to the ketogenic diet
* children suitable for surgery or parents refusing drug and diet intervention.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Epilepsy Control Response Rate | During the study period (16 weeks)
  Epilepsy control response rate: defined as an absolute reduction of ≥50% in seizure frequency at follow-up compared with baseline
  =(No attack + Marked effect + Effective)/Total number of cases × 100%.

SECONDARY OUTCOMES:
Inflammatory Marker Levels | During the study period (16 weeks)]
  This indicator aims to evaluate the effect of the ketogenic diet on the levels of inflammatory markers in the blood of children with refractory epilepsy to reveal the potential relationship between the effects of the ketogenic diet and inflammation levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat Sen Memorial Hospital， Sun Yat Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vezzani A, Maroso M, Balosso S, Sanchez MA, Bartfai T. IL-1 receptor/Toll-like receptor signaling in infection, inflammation, stress and neurodegeneration couples hyperexcitability and seizures. Brain Behav Immun. 2011 Oct;25(7):1281-9. doi: 10.1016/j.bbi.2011.03.018. Epub 2011 Apr 5. PMID 21473909
- [Background] Wirrell E, Farrell K, Whiting S. The epileptic encephalopathies of infancy and childhood. Can J Neurol Sci. 2005 Nov;32(4):409-18. doi: 10.1017/s0317167100004388. PMID 16408569
- [Background] Chen Z, Brodie MJ, Liew D, Kwan P. Treatment Outcomes in Patients With Newly Diagnosed Epilepsy Treated With Established and New Antiepileptic Drugs: A 30-Year Longitudinal Cohort Study. JAMA Neurol. 2018 Mar 1;75(3):279-286. doi: 10.1001/jamaneurol.2017.3949. PMID 29279892
- [Background] Kwan P, Arzimanoglou A, Berg AT, Brodie MJ, Allen Hauser W, Mathern G, Moshe SL, Perucca E, Wiebe S, French J. Definition of drug resistant epilepsy: consensus proposal by the ad hoc Task Force of the ILAE Commission on Therapeutic Strategies. Epilepsia. 2010 Jun;51(6):1069-77. doi: 10.1111/j.1528-1167.2009.02397.x. Epub 2009 Nov 3. PMID 19889013
- [Background] Loscher W, Potschka H, Sisodiya SM, Vezzani A. Drug Resistance in Epilepsy: Clinical Impact, Potential Mechanisms, and New Innovative Treatment Options. Pharmacol Rev. 2020 Jul;72(3):606-638. doi: 10.1124/pr.120.019539. PMID 32540959